CLINICAL TRIAL: NCT06321250
Title: An Open-label, Multicenter Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of JMKX003948 Tablets in Patients With Renal Cell Carcinoma
Brief Title: A Study of JMKX003948 Tablets in Patients With Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Collaborators: Zhejiang Hangyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JY-JM3948-101
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Renal Cell Carcinoma Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Subjects will be assigned to pre-specified dose level to determine MTD/MAD of JMKX003948. Each treatment cycle will be 21 days.
  Interventions: Drug: JMKX003948
- Dose Expansion (Experimental): Subjects will be assigned to the recommended dose level determined in dose escalation Phase. Each treatment cycle will be 21 days.
  Interventions: Drug: JMKX003948

INTERVENTIONS:
Drug: JMKX003948 — Subjects will receive JMKX003948 tablets until disease progression

SUMMARY:
This open-label Phase 1 study will evaluate the safety, tolerability, PK characteristics and preliminarily efficacy of JMKX003948 tablets in patients with renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Has the ability to understand and willingness to sign a written informed consent form.
2. Male or female from 18 years of age or older.
3. Histologically confirmed locally advanced or metastasis clear cell renal cell carcinoma.
4. Has at least one measurable lesion per RECIST v1.1.
5. Has a life expectancy of ≥ 12 weeks.
6. Adequate organ function.

Exclusion Criteria:

1. Patients with known active CNS metastases and/or cancerous meningitis.
2. Has received any type of systemic anticancer monoclonal antibodies or other immunosuppressants within 4 weeks prior to the first dose. Has received prior chemotherapy, targeted therapy, or other investigational therapy within 2 weeks prior to the first dose.
3. Has failed to recover from a ≥ grade 2 adverse event due to prior anti-tumor therapy.
4. Has impaired heart function,or clinically significant cerebrovascular and cardiovascular disease.
5. Subjects with dysphagia or known drug absorption disorders.
6. Has a history of any other malignancy within 5 years.
7. Has severe oncological complications.
8. Is currently participating in other clinical studies.
9. Subjects with be unsuitable for participation in the trial evaluated by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Number of participants with dose limiting toxicities (DLTs) | Up to 2 months
  Number of participants with DLTs
Dose Escalation: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to 2 years
  Number of participants with AEs/SAEs to characterize the safety and tolerability of JMKX003948.
Dose Expansion: Objective Response Rate (ORR) | Up to 1 year
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
maximum plasma concentration (Cmax) | Up to 1 month
  Maximum observed concentration.
maximum plasma concentration (Tmax) | Up to 1 month
  Time to reach maximum observed plasma concentration.
Duration of Response (DoR) | Up to 1 year
  DoR is defined as the time from the date of first documented CR or PR, assessed by investigator and based on RECIST v. 1.1, to the documented date of progressive disease (PD) or death, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Caancer Hospital, Beijing, China